CLINICAL TRIAL: NCT03736551
Title: Model of Intermittent Very Low Energy Diet and eXercise for Lowering BMI in Patients With CKD (MIX UP): Feasibility Study
Brief Title: Intermittent Low Energy Diet in CKD: MIX UP Feasibility Study
Acronym: MIX-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KCH17-027; 202350 (Registry Identifier: IRAS)
Record Dates: First submitted 2018-08-01; First posted 2018-11-09 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2018-07

CONDITIONS: Chronic Kidney Diseases; Obesity
Keywords: intermittent fasting; weight loss
MeSH Terms: conditions — Renal Insufficiency, Chronic; Obesity; Intermittent Fasting; Weight Loss | interventions — Diet

STUDY DESIGN:
Intervention Model Description: Parallel arm, single blinded, randomised controlled feasibility study
Who Masked: Outcomes Assessor
Masking Description: Study outcome measures performed by assessor blinded to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will involve standard care plus an intermittent modified fasting regimen consisting of a very low energy diet (600 kcal/day) on 2 consecutive days of the week, and 5 days each week on an energy restricted diet to maintain a similar overall energy deficit of 600 kcal/day across the week (5:2 diet). All dietary intake on modified fasting days will be from LighterLife foodpacks, (4 x 150 kcal portions/day presented as milkshakes, cereal bars, soups and modified meals such as spaghetti bolognese, or macaroni cheese) providing ~600 kcal/day and 100% of the RNI for vitamins and minerals.
  Interventions: Behavioral: 5:2 diet; Behavioral: Renal Weight Management Programme
- Standard Care (Active Comparator): Renal Weight management Programme - Patients will attend individual appointments with the specialist dietitian and physiotherapist once a month, for 6 months. Dietary intervention includes a standard continuous energy restricted diet aimed at reducing daily energy intake by 600 kcal/day relative to their estimated total energy expenditure (9). In addition to the dietary intervention, the programme also includes personal exercise plans, optional pharmacotherapy (orlistat at standard dose), and development of personalised dietary and exercise goals using behavioural therapy techniques and motivational interviewing.
  Interventions: Behavioral: Renal Weight Management Programme

INTERVENTIONS:
Behavioral: 5:2 diet — very low energy diet (600 kcal/day) on 2 consecutive days of the week, and 5 days each week on an energy restricted diet to maintain a similar overall energy deficit of 600 kcal/day across the week (5:2 diet)
  Arms: Intervention
Behavioral: Renal Weight Management Programme — Dietary intervention includes a standard continuous energy restricted diet aimed at reducing daily energy intake by 600 kcal/day relative to their estimated total energy expenditure. In addition to the dietary intervention, the programme also includes personal exercise plans, optional pharmacotherapy (orlistat at standard dose), and development of personalised dietary and exercise goals using behavioural therapy techniques and motivational interviewing.

SUMMARY:
This study proposes to investigate the acceptability and efficacy of intermittent VLED (5:2 diet) plus exercise, compared with the investigator's established Weight Management Programme (WMP), in obese patients with CKD, using feasibility study methodology.

Patients will be invited to participate in the parallel arm, single blinded, randomised controlled feasibility study, and randomly allocated to 1 of 2 treatments for 6 months. The experimental arm involves an intermittent modified fasting regimen consisting of VLED (600 kcal/day) on 2 consecutive days, and 5 days each week on a modified diet to maintain an overall energy deficit of 600 kcal/day across the week (5:2 diet). The control arm will be the standard renal WMP with a continuous energy restricted diet aimed at reducing daily energy intake by 600 kcal/day.

The feasibility outcomes are: recruitment rate >50%; intervention retention rate at 6 months >60%; dietary intervention compliance; and weight loss. Secondary outcomes include safety, body composition, proteinuria, lipids, blood pressure, and eating desire. Measurements will be made at baseline, midpoint, and twice at endpoint.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 years
* KDIGO defined CKD (all categories)
* BMI ≥30kg/m2
* able to provide written informed consent in English

Exclusion Criteria:

* pregnant or breastfeeding women
* conservatively managed CKD stage 5
* palliative or active treatment for cancer
* unstable chronic liver disease
* type 1 diabetes and type 2 diabetes controlled with anti-hyperglycaemic medication
* previous bariatric surgery
* unable to provide written informed consent
* significant psychiatric disorder or uncontrolled depression
* participated in a weight management drug trial in the previous 3 months
* uncontrolled epilepsy
* alcohol or substance abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Retention rate of at least 60% in the intervention group | 6 months
  Patients attending at least 80% of monthly clinic visits, including the baseline and final study visits, and remaining compliant with the 2 consecutive days VLED throughout the 6 month intervention will be considered "completers" and count as being retained in the intervention group at 6 months.
Number of Adverse Events following intermittent very low energy diet | 6 months
  record of all adverse events including but not limited to nausea, constipation and/or diarrhoea, dehydration, hypoglycaemia, lethargy & fatigue, headaches, gallstones and gout.

SECONDARY OUTCOMES:
Recruitment rate of at least 50% of potential participants meeting inclusion and exclusion criteria | 1 year
  at least 50% of those meeting the referral criteria and are approached to participant, consent to participating in the study
Compliance with dietary intervention from dietary records | 6 months
  at least 70% compliance with prescribed diet
Weight change (kg) | 6 months
  change in weight from baseline to 6 months
kidney function (eGFR ml/min CKD EPI equation) | 6 months
  monitoring if estimated kidney function declines during the study or if symptomatic for dehydration.
Waist circumference (cm) | 6 months
  change in waist circumference measured in cm at level of umbilicus
Body composition | 6 months
  lean and fat mass (kg) estimated by bioelectrical impedance analysis
Exercise capacity - 6 minute timed walk test | 6 months
  distance walked (m) in 6 minutes
Exercise capacity - sit to stand 60 | 6 months
  number (count) of sit to stand movements in 60 seconds
Proteinuria | 6 months
  urinary protein to creatinine ratio
Total Cholesterol | 6 months
  plasma total cholesterol concentration
Triglycerides | 6 months
  plasma triglycerides concentration
LDL cholesterol | 6 months
  plasma LDL cholesterol concentration
HDL cholesterol | 6 months
  plasma HDL cholesterol concentration

CONTACTS AND LOCATIONS:
Overall Officials: Helen L MacLaughlin, PhD, Principal Investigator — King's College Hospital NHS Fundation Trust
Locations (1):
- King's College Hospital, London, United Kingdom